CLINICAL TRIAL: NCT01667926
Title: Randomized, Double-blind Ketamine Augmentation in Chronically Suicidal, Treatment-resistant Major Depression
Brief Title: Ketamine Versus Placebo for Treatment Resistant Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Cristina Cusin, MD, Instructor HSM, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012-P-001042
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine (Experimental): Subject will receive 6 infusions of ketamine over three weeks.
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): Subjects will receive 6 infusions of normal saline over 3 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — ketamine infusions twice a week for three weeks, total of 6 infusions as augmentation of ongoing antidepressant regimen.
  Arms: Ketamine
Drug: Placebo
  Arms: Placebo

SUMMARY:
Ketamine infusions resulted in an acute reduction in global depression scores and in severity of suicidal ideation. The investigators therefore plan to investigate the feasibility and efficacy of repeated intravenous administration of ketamine in severely depressed, treatment resistant patients. The results of the study could lead to development of new strategies for treating depression.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient with sever treatment resistant depression
* Currently depressed
* Currently under regular psychiatric care
* On an aggressive antidepressant regimen, stable for 4 weeks.

Exclusion Criteria:

* No history of other major psychiatric illness, including bipolar
* No history of psychosis
* No history of drug abuse
* No major medical illness or unstable medical problem

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-01; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Cusin, M.D., Principal Investigator — MGH Department of Psychiatry
Locations (1):
- Depression Clinical and Reseach Program - MGH, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatients were recruited primarily through referrals.
Groups:
- Placebo: Subjects will receive 6 infusions of normal saline over 3 weeks.
  Placebo
- Screen Fail/No Baseline: Participants who signed informed consent and were screened but did not meet study inclusion/exclusion criteria.
  Participants in the screen fail group were not randomized to either Ketamine nor placebo and did not receive any infusions.
Period: Overall Study
Arm/Group | Ketamine | Placebo | Screen Fail/No Baseline
Started | 13 | 13 | 11
Completed | 8 | 9 | 0 (Participants in the screen fail group were not randomized in the study.)
Not Completed | 5 | 4 | 11
Not completed — Withdrawal by Subject | 1 | 2 | 2
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Time committment | 0 | 0 | 2
Not completed — Inclusion/Exclusion Criteria | 0 | 0 | 5
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Side effects | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Placebo | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (13.6) | 45.3 (11.7) | 45.4 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 6 | 10 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale - Suicidal Ideation (HDRS-SI)
Description: The HDRS-SI score consists of a single item on the Hamilton Depression Rating Scale (HDRS). Scores range from 0 to 4, with 0 representing no suicidal ideation, and 4 representing a suicide attempt.
Time Frame: up to 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 8 | 9
units on a scale | 1.6 (1.4) | 1.6 (1.4)

2. Secondary Outcome: HDRS-28 Total
Description: Hamilton Depression Rating Scale Total scores after completing 6 infusions. Scores may range from 0-81 with higher scores indicating greater depression severity. HDRS-28 score ≤ 7 was considered remission.
Time Frame: up to 5 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 8 | 9
units on a scale | 20.2 (11.1) | 20.0 (10.7)

ADVERSE EVENTS:
Time Frame: up to 3 months
Description: Adverse events were tracked from Baseline to three months after final infusion in a naturalistic "follow-up" phase.
Arm/Group | Ketamine | Placebo
Serious Adverse Events (participants affected / at risk) | 2/13 | 0/13
Other Adverse Events (participants affected / at risk) | 3/13 | 1/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=13) | Placebo (N=13)
Unrelated hospitalization (Infections and infestations) | 1 (1) | 0 (0) — The subject was hospitalized due to syncope. This event very unlikely related to the study medication, due to the significant time delay between the final infusion and the episodes of syncope. The most probable explanation is a viral infection.
Worsening Depression (Psychiatric disorders) | 2 (2) | 0 (0) — Participant was hospitalized due to worsening depression and suicidal ideation. Study team was notified by the participant via phone call or email.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=13) | Placebo (N=13)
Ketamine side effects (General disorders) | 2 (3) | 0 (0) — Including dizziness, fever, fainting, and detachment from reality
Psychiatric Hospitalization (Psychiatric disorders) | 0 (0) | 1 (1)
Diarrhea (General disorders) | 1 (1) | 0 (0)
Blood Pressure elevated (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No